CLINICAL TRIAL: NCT03926975
Title: The Effect of a Scleral Lens on the Anterior Chamber Depth and Minimum Rim Width
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, MKWalker, Lecturer, University of Houston
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000747
Record Dates: First submitted 2019-04-18; First posted 2019-04-25 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Subjects are all non-scleral lens wearers. One eye (test) will be selected to wear a scleral lens, and the contralateral eye (control) will not wear any lens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental: Scleral Lens (Experimental): One eye will be randomly selected to wear a scleral lens for a 6-hour testing period.
  Interventions: Device: Scleral Lens
- Control: no lens (Active Comparator): The contralateral eye will not wear a lens.
  Interventions: Other: No lens

INTERVENTIONS:
Device: Scleral Lens — The contact lens will be worn on one eye.
  Arms: Experimental: Scleral Lens
Other: No lens — No lens worn on the contralateral control eye
  Arms: Control: no lens

SUMMARY:
The purpose of this study is to evaluate the use of two instruments to measure changes in two ocular structures: 1) the anterior chamber depth (ACD) - measured using low coherence optical biometry, and 2) minimum rim width of the optic nerve head (MRW) - measured using optical coherence tomography. Changes in these ocular structures indicate fluctuations in intraocular pressure (IOP) and will be measured during scleral contact lens (SGP) wear to determine if SGP wear influences IOP. We hypothesize that a scleral lens increases the intraocular pressure (IOP) during active wear and that the ACD and MRW will also change.

DETAILED DESCRIPTION:
Contact lenses are often used to correct vision blur. The most common types of contact lenses include those referred to as 'soft' and 'rigid'. Visual acuity through rigid lenses often surpasses that of soft lenses. Historically, these lenses have been small in diameter, and hence patients also felt discomfort when wearing the lenses. Scleral lenses are relatively new, customized devices that have gained popularity with patients and practitioners in the past 5-10 years, because they are more comfortable and provide more stable vision than the small diameter rigid contact lenses. However, relatively little is known about the physiologic response of the eye to the scleral lens, or the long-term effects of their use, since they are such a new modality.

Maintaining the IOP within the eye is imperative to prevent damage to ocular tissue, which can occur in glaucoma. Given the landing of scleral lens overlying the sclera and ciliary body, which assist in modulating the transport of fluid in the eye, there is a potential for these lenses to impinge on fluid drainage which could lead to increases of IOP during scleral lens wear. The placement of the lens creates an obstacle in evaluating IOP while the lens is actually on the eye (covering the cornea), and since increases in IOP may only occur during lens wear, which is removed when determining clinical IOP measurements, it is difficult to monitor IOP during scleral lens wear with traditional IOP instrumentation (ie. iCare, Goldman, etc).

Optical coherence tomography is a non-invasive imaging technology that has revolutionized how the retina and optic nerve are clinically evaluated. The optic nerve head is typically assessed using radial scans, from which the minimal distance from the Bruch's membrane opening to the inner limiting lamina is quantified as the minimum rim width (MRW). With changes in IOP, the MRW is known to also change in thickness. Many studies are investigating the MRW changes during IOP fluctuations, with studies finding a decrease in MRW during acute IOP increase. In this project, MRW will be used to indirectly assess changes in IOP by measuring the MRW periodically during active scleral lens wear.

In addition, we are incorporating low coherence optical biometry (Lenstar) to evaluate the effect of the scleral lens pressure on the anterior chamber. Using the Lenstar, corneal thickness, anterior chamber depth (ACD), lens thickness and vitreous chamber depth can be quantified. In this project, ACD will be used to indirectly evaluate changes in the pressure within the anterior chamber. The assumption is that the ACD will change based on changes in pressure in the scleral lens tear reservoir.

This study will add to the knowledge of how the scleral lens affects the dynamic pressure system of the eye. Based on the implications for disease with chronic increases and fluctuations in IOP, this is important information to understand with the scleral lens, a relatively new refractive treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* young, normal individuals

Exclusion Criteria:

* IOP > 20mm in either eye, and h/o ocular hypertension, glaucoma, or ocular surgery that can affect IOP.
* h/o scleral lens wear or current scleral lens wear

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in minimum rim width from baseline to 6-hours SL wear | at baseline, after 2-hours lens wear, and after 6-hours lens wear
  The Bruch's membrane opening to the inner limiting lamina (termed the minimum rim width) will be measured at the optic nerve head.

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | at baseline, after 2-hours lens wear, and after 6-hours lens wear
  IOP will be measured using the Diaton and iCare tonometers
Anterior Chamber Depth (ACD) | at baseline, after 2-hours lens wear, and after 6-hours lens wear
  ACD will be measured with the Lenstar A-scan

CONTACTS AND LOCATIONS:
Overall Officials: Maria Walker, Principal Investigator — University of Houston
Locations (1):
- University Eye Institute, Houston, Texas, United States

REFERENCES:
- [Derived] Walker MK, Pardon LP, Redfern R, Patel N. IOP and Optic Nerve Head Morphology during Scleral Lens Wear. Optom Vis Sci. 2020 Sep;97(9):661-668. doi: 10.1097/OPX.0000000000001567. PMID 32932395